CLINICAL TRIAL: NCT03989245
Title: Measuring the Impact of Care in the Cognitive Behavioural Unit
Acronym: IMPACTUCC
Status: Recruiting | Type: Observational
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A02869-46
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Severe Disruptive Behaviour Disorders
Keywords: Severe disruptive behaviour disorders; Cognitive Behavioural Unit; Geriatric Follow-up and Rehabilitation Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Target arm: UCC (Cognitive Behavioural Unit): Patients receiving care in Cognitive Behavioural Unit (UCC )
- Control arm: SSR (Geriatric Follow-up and Rehabilitation Unit): Patients receiving care in Geriatric Follow-up and Rehabilitation Care Unit (SSR)

SUMMARY:
The purpose of this study is to compare the rate of re-hospitalizations in relation to a disruptive behaviour disorder (at 3 and 6 months) between patients who have received care in Cognitive Behavioural Unity (UCC ) and those who have received care in Geriatric Follow-up and Rehabilitation Care Unit (SSR).

DETAILED DESCRIPTION:
The purpose of this muliticentric non-interventional study is to compare the rate of re-hospitalization in relation to a disruptive behaviour disorder between patients receiving care in Cognitive Behavioural Unity UCC (target arm) and those who have received care in Geriatric Care Unit and Rehabilitation SSR (Control arm ).

At Inclusion (Month 0) : Inclusion of patients admitted in UCC or in geriatric SSR units for less than 8 days after obtaining of their non opposition.

Following data: Socio-educational Level, somatic and psychiatric comorbidities, classification of the type of dementia, evolution of nutritional status, biology (hemoglobin, creatinine, albuminemia), cognitive evaluation, treatment, pain assessment, assessment of disruptive behaviour disorders, discharge modalities, assistance plan, legal protection (before and after hospitalization), types of restraints, measurement of fall rates and their consequences, pathology and/or symptoms observed ( incidents) during hospitalization and vital status will be collected at inclusion and follow-up (1, 3 and 6 months ).

At 1 month (M1), exit from hospitalization (M1): Data provided by Investigator .

At 3 months (M3) and 6 months (M6) after discharge from hospital in UCC or SSR: Sponsor's Clinical Research Associateall call patient (or his legal representative) or to the primary caregiver or attending physician or EHPAD coordinating physician for collection of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* 70 ≥ years of age
* Patient with severe disruptive behaviour disorders with a score (Frequency X Severity) >7 to at least one of the 7 items targeted on Clinician Neuropsychaitric Inventury (NPI-Es) scale
* Patient who was not cared for in Cognitive Behavioural Unit (UCC) within 6 months prior to admission
* Patient entered center less than 8 days
* Affiliation to a social security scheme
* Patient or legal representative has expressed his non-opposition

Exclusion Criteria:

* 70 < years of age
* Patient with no score (FXG) >7 to at least one of the 7 items targeted on Clinician Neuropsychaitric Inventury NPI-ES scale
* Patient who was cared for in UCC within 6 months of admission
* Entered Centre for 8 days or more
* Not affiliated or entitled to a social security scheme
* Patient or legal representative has expressed his opposition

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients receiving care in Cognitive Behavioural Unit (UCC ) and Geriatric Follow-up and Rehabilitation Unit (SSR)
Sampling Method: Non-Probability Sample
Enrollment: 588 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Compare the rate of re-hospitalizations in relation to a disruptive behaviour disorder according Clinician Neuropsychaitric Inventury (NPI-Es) scaleaccording | 6 months

SECONDARY OUTCOMES:
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) score | 6 months
Screening for a nutritional disorder according Body Mass Index (BMI) score | 1 month
Assessment of somatic-comorbidities according Charlson scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Drunat, MD, Study Chair — Psychiatric Geriatric Department, Bretonneau hospital
Locations (1):
- Psychiatric Geriatric Department, Bretonneau hospital, Paris, Île-de-France Region, France